CLINICAL TRIAL: NCT03867773
Title: Time Restricted Feeding (4-hour Versus 6-hour) for Weight Loss in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1525
Record Dates: First submitted 2019-03-04; First posted 2019-03-08 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-hour Time restricted feeding (Experimental): 4-h TRF subjects will consume food ad libitum between 3pm and 7pm (4-h feeding window), and refrain from eating and drinking caloric beverages from 7pm to 3pm (20-h fasting window) each day. These subjects will not be instructed to limit/monitor energy intake during the feeding window. Subjects will be encouraged to drink plenty of water during the fasting period.
  Interventions: Behavioral: Time restricted feeding
- Control (No Intervention): Controls will be instructed to maintain their weight throughout the trial, and not to change eating or physical activity habits. Controls will visit the research center at the same frequency as the TRF groups (for outcome measurements).
- 6-hour Time restricted feeding (Experimental): 6-h TRF subjects will consume food ad libitum between 1pm and 7pm (6-h feeding window), and refrain from eating and drinking caloric beverages from 7pm to 1pm (18-h fasting window) each day. These subjects will not be instructed to limit/monitor energy intake during the feeding window. Subjects will be encouraged to drink plenty of water during the fasting period.
  Interventions: Behavioral: Time restricted feeding

INTERVENTIONS:
Behavioral: Time restricted feeding — TRF subjects will consume food ad libitum during the feeding window (4-h or 6-h window), and refrain from eating during the fasting window (20-h or 18-h window)
  Arms: 4-hour Time restricted feeding; 6-hour Time restricted feeding

SUMMARY:
The aims of this proposal are to compare the effects of 4-h versus 6-h time restricted feeding (TRF) on body weight and metabolic disease risk factors in adults with obesity. To test the study objectives, a 10-week randomized, controlled, parallel-arm trial, divided into 2 consecutive periods: (1) 2-week baseline period; and (2) 8-week TRF weight loss period, will be implemented. Obese subjects will be randomized to 1 of 3 groups: (1) 4-h TRF, (2) 6-h TRF, or a no-intervention control group. This study will be the first randomized controlled trial to compare 4-h versus 6-h TRF.

DETAILED DESCRIPTION:
Modest weight loss of 5-10% is sufficient to reduce metabolic disease risk in obese individuals. The first line of therapy prescribed for weight loss is daily calorie restriction (CR; 25% restriction every day). However, adherence to CR greatly diminishes after 4-6 weeks, due to subject frustration with constantly having to count calories and never being able to eat freely. In light of these issues with CR, another approach that limits timing of food intake, instead of number of calories consumed, has been developed. This strategy is termed time restricted feeding (TRF), and involves confining the period of food intake to 8 h/d (10 am to 6 pm) without calorie counting. Preliminary findings of 8-h TRF demonstrate modest weight loss and blood pressure reductions after 12 weeks. What remains unknown however, is whether shorter feeding windows during TRF (such as 4-h or 6-h feeding windows) can produce even greater weight loss in obese adults. Also of interest, is the impact of these shorter feeding windows on metabolic disease risk indicators (such as plasma lipids, blood pressure, and insulin resistance, inflammation and oxidative stress). Accordingly, the aims of this proposal are: AIM 1: To compare the effects of 4-h versus 6-h time restricted feeding (TRF) on body weight in adults with obesity; AIM 2: To compare the effects of 4-h versus 6-h TRF on metabolic disease risk factors in adults with obesity. To test the study objectives, a 10-week randomized, controlled, parallel-arm trial, divided into 2 consecutive periods: (1) 2-week baseline period; and (2) 8-week TRF weight loss period, will be implemented. Obese subjects will be randomized to 1 of 3 groups: (1) 4-h TRF, (2) 6-h TRF, or a no-intervention control group. This study will be the first randomized controlled trial to compare 4-h versus 6-h TRF on body weight and metabolic disease risk markers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* body mass index (BMI) between 30.0 and 49.9 kg/m2;
* age between 18 and 65 years; sedentary (light exercise less than 1 h per week) or moderately active (moderate exercise 1 to 2 h per week);
* weight stable for >3 months prior to the beginning of the study (gain or loss <4 kg);
* able to give written informed consent

Exclusion Criteria:

* Smoker; diabetic;
* taking weight loss medications;
* taking medication that requires eating food before (or with) the medication; history of eating disorders;
* night-shift workers;
* perimenopausal;
* pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 in body weight | Measured at week 1 and 8
  Measured by an electronic scale

SECONDARY OUTCOMES:
Change from baseline to week 8 in body composition | Measured at week 1 and 8
  Measured by DXA
Change from baseline to week 8 in Insulin resistance | Measured at week 1 and 8
  Measured as HOMA-IR
Change from baseline to week 8 in Fasting glucose | Measured at week 1 and 8
  Measured with a hexokinase reagent kit
Change from baseline to week 8 in Fasting insulin | Measured at week 1 and 8
  Measured as total immunoreactive insulin
Change from baseline to week 8 in Blood pressure | Measured at week 1 and 8
  Measured by a blood pressure cuff
Change from baseline to week 8 in adverse events | Measured weekly from baseline to week 8
  Measured by questionnaire
Change from baseline to week 8 in plasma lipids | Measured at week 1 and 8
  Measured by outside lab (Medstart, IN)
Change from baseline to week 8 in heart rate | Measured at week 1 and 8
  Measured by a blood pressure cuff
Change from baseline to week 8 in inflammatory markers (TNF-a, IL-6) | Measured at week 1 and 8
  Measured by ELISA
Change from baseline to week 8 in oxidative stress (8-isoprostane) | Measured at week 1 and 8
  Measured by ELISA
Change from baseline to week 8 in calorie and macronutrient intake | Measured at week 1 and 8
  Measured by food record
Change from baseline to week 8 in physical activity (steps/d) | Measured at week 1 and 8
  Measured by activity monitor
Change from baseline to week 8 in diet adherence | Measured weekly from baseline to week 8
  Measured by a questionnaire
Change from baseline to week 8 in sleep quality | Measured at week 1 and 8
  Measured by a questionnaire
Change from baseline to week 8 in insomnia severity | Measured at week 1 and 8
  Measured by a questionnaire
Change from baseline to week 8 in risk of sleep apnea | Measured at week 1 and 8
  Measured by a questionnaire
Change from baseline to week 8 in sex steroid levels (estrogen, androgens, sex hormone binding globulin) | Measured at week 1 and 8
  Measured by a ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cienfuegos S, Gabel K, Kalam F, Ezpeleta M, Lin S, Varady KA. Changes in body weight and metabolic risk during time restricted feeding in premenopausal versus postmenopausal women. Exp Gerontol. 2021 Oct 15;154:111545. doi: 10.1016/j.exger.2021.111545. Epub 2021 Aug 31. PMID 34478825
- [Derived] Cienfuegos S, Gabel K, Kalam F, Ezpeleta M, Wiseman E, Pavlou V, Lin S, Oliveira ML, Varady KA. Effects of 4- and 6-h Time-Restricted Feeding on Weight and Cardiometabolic Health: A Randomized Controlled Trial in Adults with Obesity. Cell Metab. 2020 Sep 1;32(3):366-378.e3. doi: 10.1016/j.cmet.2020.06.018. Epub 2020 Jul 15. PMID 32673591